CLINICAL TRIAL: NCT03629431
Title: Multicenter, Randomized, Open Study, Assessing Prophylactic Noninvasive Ventilation in Intensive Care Unit vs Postoperative Standard Care for Patients With High Risk of Postoperative Pulmonary Complication With Preoperative ARISCAT Score
Brief Title: Prophylactic Noninvasive Ventilation in vs Postoperative Standard Care in High Risk Patients According to ARISCAT Score
Acronym: ANTICIPUSC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Cancerologie de l'Ouest (Other)
Collaborators: Direction Générale de l'Offre de Soins (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ICO-A-2016-04
Record Dates: First submitted 2018-07-03; First posted 2018-08-14 (Actual); Results first posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2020-03

CONDITIONS: Surgical Patients; Pulmonary Complication
Keywords: ARISCAT; complications; postoperative

STUDY DESIGN:
Intervention Model Description: This is a study phase III, multicentre, comparative, randomized, controlled, superiority and open
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- postoperative standard care (Active Comparator): Standard care after surgery in postoperative unit
  Interventions: Procedure: postoperative standard care
- Prophylactic non-invasive ventilation (Experimental): Prophylactic noninvasive ventilation in postoperative and intensive care unit
  Interventions: Procedure: Prophylactic non-invasive ventilation

INTERVENTIONS:
Procedure: Prophylactic non-invasive ventilation — The sessions of NIV last 1 hour and are repeated every 2 to 3 hours with a goal of a daily assistance period of 6 to 8 hours for a minimum of 24 hours.
  The sessions are spaced by periods of unassisted ventilation of 2 hours allowing the patient to rest, feed, receive care including physiotherapy sessions.
  Arms: Prophylactic non-invasive ventilation
Procedure: postoperative standard care — Standard care received postoperatively
  Arms: postoperative standard care

SUMMARY:
Postoperative pulmonary complications are one of the most common complications after surgery.

Noninvasive ventilation has been proposed post-operatively to prevent postoperative pulmonary complications.

Prophylactic noninvasive ventilation performed systematically in a non-specific population is without interest.

The difficulty for the practitioner is to target patients at higher risk of developing a postoperative pulmonary complications in order to guiding them to a post-operative specialized care pathway.

The use of the ARISCAT score, validated on a large European prospective cohort, makes it possible to evaluate, preoperatively, the risk of occurrence of postoperative pulmonary complication in the patient.

The hypothesis of the present research is that early postoperative preventive treatment with noninvasive ventilation, in patients at risk of postoperative pulmonary complications according to the preoperative evaluation according to the ARISCAT score, could have an interest in reducing these complications with a superior efficiency over standard techniques.

DETAILED DESCRIPTION:
After verification of eligibility criteria and ARISCAT score, patients at high risk of COPD are randomized in the study.

At the exit of the operating room, patients are referred to the services according to their randomization arm :

* arm with prophylactic noninvasive ventilation in intensive care unit. Patients will receive noninvasive ventilation for a maximum of 48 hours. Sessions last 1 hour and are repeated every 2 to 3 hours
* arm with standard care in conventional care unit. Patients receive standard care such as physiotherapy.

In both arms, patient follow-up is 7 days maximum.

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years of age or older
* Patient scheduled for surgery or considered semi-urgent (=pre-anesthesia consultation <48h before the surgical procedure) under General Anesthesia or under Loco-Regional Anesthesia
* Patient with an ARISCAT score higher than or equal to 45 - Obtaining the signed written consent of the patient
* Patient affiliated to a social security scheme

Exclusion Criteria:

* Minor patients, pregnant or lactating women
* Obstetrical interventions
* Surgery under Local Anesthesia or Peripheral Nerve,
* Interventions taking place outside an interventional room
* Interventions for previous surgical complications
* Second surgery during study
* Organ transplantation
* Patients already intubated in preoperative
* Outpatient surgery
* Refusal of participation or inability to issue informed consent
* Person deprived of liberty or adult under guardianship
* Participation in another interventional study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2017-11-03 (Actual); Primary Completion 2019-10-16 (Actual); Study Completion 2019-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: DENIS DUPOIRON, MD, Principal Investigator — Institut de Cancérologie de l'Ouest
Locations (3):
- France (3):
  - Chu D'Angers, Angers
  - Institut de Cancerologie de L'Ouest, Angers
  - Ch Du Mans, Le Mans

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abrard S, Rineau E, Seegers V, Lebrec N, Sargentini C, Jeanneteau A, Longeau E, Caron S, Callahan JC, Chudeau N, Beloncle F, Lasocki S, Dupoiron D. Postoperative prophylactic intermittent noninvasive ventilation versus usual postoperative care for patients at high risk of pulmonary complications: a multicentre randomised trial. Br J Anaesth. 2023 Jan;130(1):e160-e168. doi: 10.1016/j.bja.2021.11.033. Epub 2022 Jan 5. PMID 34996593

RESULTS

PARTICIPANT FLOW:
Groups:
- Prophylactic Non-invasive Ventilation: Prophylactic noninvasive ventilation in postoperative and intensive care unit
  Prophylactic non-invasive ventilation: The sessions of NIV last 1 hour and are repeated every 2 to 3 hours with a goal of a daily assistance period of 6 to 8 hours for a minimum of 24 hours.
  The sessions are spaced by periods of unassisted ventilation of 2 hours allowing the patient to rest, feed, receive care including physiotherapy sessions.
Period: Overall Study
Arm/Group | Postoperative Standard Care | Prophylactic Non-invasive Ventilation
Started | 133 | 133
Completed | 128 | 125
Not Completed | 5 | 8
Not completed — Withdrawal by Subject | 5 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Postoperative Standard Care | Prophylactic Non-invasive Ventilation | Total
Number analyzed (Participants) | 128 | 125 | 253
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.8 (11.3) | 68.10 (9.6) | 67.4 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 27 | 50
  Male | 105 | 98 | 203
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Acute Respiratory Failure Within the First 7 Days Following Surgery (or Until Hospital Discharge if Occurring First)
Description: The outcome was reported as the count of participants who experienced acute respiratory failure, defined as the need for invasive or non-invasive mechanical ventilation within 7 days after surgery or until hospital discharge, whichever occurred first. All events were validated by an adjudication committee in this randomized, single-blind trial.
Time Frame: Up to 7 days post-surgery or until hospital discharge (study duration: 23 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Postoperative Standard Care | Prophylactic Non-invasive Ventilation
Number analyzed (Participants) | 128 | 125
Participants | 35 | 30

2. Secondary Outcome: Number of Participants With Healthcare-Associated Infections Within 30 Days After Surgery (Defined According to CDC Criteria)
Description: The outcome was reported as the count of participants who developed healthcare-associated infections within 30 days after surgery, defined according to the Centers for Disease Control and Prevention (CDC) criteria. All events were validated by an adjudication committee
Time Frame: 30days
Measure: Count of Participants; unit: Participants
Arm/Group | Postoperative Standard Care | Prophylactic Non-invasive Ventilation
Number analyzed (Participants) | 128 | 125
Participants
  Pleural effusion | 41 | 36
  Bronchospasm | 0 | 3
  Atelectasis | 73 | 61
  Upper airways obstruction | 10 | 4
  Pulmonary edema | 15 | 11
  Aspiration pneumonitis | 1 | 2
  Respiratory infection | 3 | 3
  Pneumothorax | 4 | 6

3. Secondary Outcome: Reintubation Rate Within 7 Days
Description: Number of patients reintubated
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Postoperative Standard Care | Prophylactic Non-invasive Ventilation
Number analyzed (Participants) | 128 | 125
Participants | 8 | 9

ADVERSE EVENTS:
Time Frame: From signature of consent to the end of follow up (30 days)
Arm/Group | Postoperative Standard Care | Prophylactic Non-invasive Ventilation
All-Cause Mortality (participants affected / at risk) | 2/128 | 3/125
Serious Adverse Events (participants affected / at risk) | 19/128 | 15/125
Other Adverse Events (participants affected / at risk) | 128/128 | 125/125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Postoperative Standard Care (N=128) | Prophylactic Non-invasive Ventilation (N=125)
Acute Renal Failure (Renal and urinary disorders) | 2 (2) | 2 (2)
Transient ischemic attack (Nervous system disorders) | 1 (1) | 0
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1)
Stroke (Nervous system disorders) | 1 (1) | 1 (1)
cardiogenic shock (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0
cholecystisis (Hepatobiliary disorders) | 0 | 1 (1)
Convulsive seizure (Psychiatric disorders) | 0 | 1 (1)
Hemodynamic failure (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Cardiac rythm disorders (Cardiac disorders) | 1 (1) | 0
bronchail congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0
Pericardial effusion (Blood and lymphatic system disorders) | 1 (1) | 0
Ileus (Gastrointestinal disorders) | 0 | 2 (2)
Inhalation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0
food intolerance (General disorders) | 1 (1) | 0
mediastinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0
pneumopathy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1)
Bleeding (Blood and lymphatic system disorders) | 2 (2) | 3 (3)
Multiple organ failure (General disorders) | 1 (1) | 1 (1)
Bowel obstruction (Gastrointestinal disorders) | 1 (1) | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Postoperative Standard Care (N=128) | Prophylactic Non-invasive Ventilation (N=125)
chirurgical complication (General disorders) | 17 (17) | 7 (7)
Cardiovascular disorders (Cardiac disorders) | 61 (74) | 66 (67)
Multiple organ failure (General disorders) | 44 (52) | 31 (37)
Digestive disorders (Gastrointestinal disorders) | 46 (55) | 52 (58)
psycahtric disorders (Psychiatric disorders) | 23 (26) | 25 (28)
Infection (Infections and infestations) | 49 (55) | 33 (37)
Complications of non-invasive ventilation (General disorders) | 31 (33) | 54 (69)
Postoperative Pulmonary Complication (Respiratory, thoracic and mediastinal disorders) | 87 (147) | 79 (126)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-19): https://cdn.clinicaltrials.gov/large-docs/31/NCT03629431/Prot_SAP_000.pdf